CLINICAL TRIAL: NCT06523426
Title: Evaluation of Ambulatory Endoscopic Spinal Surgery in the Geriatric Population
Brief Title: Ambulatory Geriatric Endoscopic Spine
Acronym: AGES
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/92
Record Dates: First submitted 2024-07-09; First posted 2024-07-26 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Decompression
Keywords: outpatient surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient treated by spinal endoscopy: elderly patients, over 75 years old, treated by spinal endoscopy
  Interventions: Diagnostic Test: Patient treated by spinal endoscopy

INTERVENTIONS:
Diagnostic Test: Patient treated by spinal endoscopy — Questionnaire administered by surgeon; assessment of level of autonomy for activities of daily living

SUMMARY:
The research focuses on evaluating the clinical outcomes of endoscopic lumbar decompression surgery performed in an outpatient setting for patients over 75 years old. This prospective, multicentric, non-interventional study aims to assess the feasibility and effectiveness of endoscopic techniques, specifically biportal and uniportal approaches, in reducing operative morbidity and hospital stay duration within this demographic. The primary objective is to determine the success rate of outpatient treatment using these endoscopic procedures in elderly patients

DETAILED DESCRIPTION:
This study investigates the clinical outcomes of endoscopic lumbar decompression surgery performed in an outpatient setting for patients over 75 years old. Given the increasing prevalence of spinal pathologies in aging populations, traditional surgical approaches pose significant morbidity and extended hospital stays, especially for the elderly. Recent advancements in less invasive endoscopic techniques offer promising alternatives that may reduce these risks. This prospective, multicentric, non-interventional study aims to evaluate the feasibility and effectiveness of endoscopic lumbar decompression, specifically biportal and uniportal approaches, in reducing operative morbidity and hospital stay duration within this demographic.

Scientific Justification Spinal pathologies, particularly degenerative conditions of the lumbar spine, are common and lead to significant healthcare costs. With the aging population in developed countries, the incidence of these pathologies is increasing, with 100% of individuals over 60 years old showing structural degenerative changes and 60% experiencing related symptoms. Current surgical treatments, such as conventional lumbar decompression, often result in prolonged hospital stays and high morbidity, particularly among the elderly who typically present with multiple comorbidities, increased bone fragility, and functional limitations. Endoscopic surgery, a less invasive alternative, has demonstrated excellent outcomes in recent studies, including lower complication rates and shorter recovery times. However, its effectiveness in the outpatient setting for the geriatric population remains unstudied.

Treatment/Strategy/Procedure The study involves endoscopic lumbar decompression surgery, utilizing either biportal or uniportal techniques, performed on patients over 75 years old in an outpatient setting. This approach aims to minimize surgical trauma and preserve the physiological function and stability of the lumbar spine.

Follow-Up Patients will be followed for three months post-surgery to monitor clinical improvements and identify any peri- or post-operative complications. Data collected will include clinical examinations, quality of life assessments, medical history, ongoing treatments, and responses to self-administered questionnaires. The follow-up visit at three months will gather comprehensive information on patient progress, including clinical examinations, imaging data, therapeutic interventions, and medication use.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 75 years.
* Patient consulting for a medical condition involving a spinal pathology at the center, for which endoscopic lumbar decompression on one level is indicated.

Exclusion Criteria:

* Patients under guardianship or trusteeship.
* Individuals deprived of liberty by judicial or administrative decision.
* Individuals undergoing psychiatric treatment under constraint requiring consent from a legal representative.
* Individuals admitted to a health or social institution for purposes other than research.
* Individuals unable to give consent.
* Individuals under legal protection.
* Patients not affiliated with a social security system.
* Patients suffering from infectious, traumatic, or tumoral spinal pathology.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient for whom an indication for ambulatory endoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Success of outpatient care : Number of patient with convention hospitalization or readmission after endoscopic surgery | 3 months visit
  The success of ambulatory management is the number of patients for whom an indication for endoscopic surgery is given and performed without the need for conventional hospitalization secondary to surgery, or readmission within 30 days of surgery

SECONDARY OUTCOMES:
Evaluation of Treatment Efficacy | Inclusion visit, 3 months visit
  Evolution of perceived health scores specific to the treated pathology. ODI (Oswestry Disability Index) is a self-questionnaire with 10 items. Each question is rated from 0 to 5 and total score that varies from 0 to 50
Evaluation of Treatment Safety | Inclusion visit, 3 months visit
  Number of serious medical complications
Evaluation of Treatment Safety | Inclusion visit, 3 months visit
  Number of surgical site infections.
Evaluation of Treatment Safety | Inclusion visit, 3 months visit
  Number of mechanical complications.
Evaluation of Treatment Safety | Inclusion visit, 3 months visit
  Number of neurological complications.
Evaluation of Treatment Safety | Inclusion visit, 3 months visit
  Number of surgical re-interventions.
Evaluation of Treatment Efficacy | Inclusion visit, 3 months visit
  Evaluation of quality of life by self-questionnaire EQ-5D-5L
Evaluation of Treatment Efficacy | Inclusion visit, 3 months visit
  Evaluation of geriatric autonomy by IADL.
Evaluation of Treatment Efficacy | Inclusion visit, 3 months visit
  Evaluation of quality of life by self-questionnaire ODI
Evaluation of Treatment Efficacy | Inclusion visit, 3 months visit
  Evaluation of quality of life by self-questionnaire SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BOUYER, PROF, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- France (3):
  - CHU DE Bordeaux, Bordeaux
  - Cliniques Terrefort Bordeaux-Bruges, Bruges
  - Clinique Saint Jean - Sud de France, Saint-Jean-de-Védas